CLINICAL TRIAL: NCT00692146
Title: A Double-Blind, Randomized, Single-Centre, Placebo-Controlled, Crossover Study to Investigate the Effects of a Single Oral Dose of AZD1386 on Intradermal Capsaicin Evoked Pain Symptoms and Heat Sensitivity in Healthy Volunteers
Brief Title: Study to Investigate the Effects Single Oral Dose of AZD1386 (Capsaicin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD Medical Science Director, AstraZeneca R&D Södertälje
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5090C00009
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Capsaicin Evoked Pain; Heat Sensitivity
Keywords: Proof of Mechanism; Capsaicin evoked pain
MeSH Terms: interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 36 subjects receiving a specified volume of the active component AZD1386 in a single dose.
  Interventions: Drug: AZD1386
- 2 (Placebo Comparator): 36 subjects receiving a specified volume of placebo in a single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — Oral solution fixed dose (95 mg given orally on two occasions)
  Arms: 1
Drug: Placebo — Oral solution fixed dose (95 mg given orally on two occasions)
  Arms: 2

SUMMARY:
A double-blind, randomized, single-centre, placebo-controlled, crossover study to investigate the effects of a single oral dose of AZD1386 on intradermal capsaicin evoked pain symptoms and heat sensitivity in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Clinical normal physical findings, including BP, pulse rate >45 bpm, ECG and laboratory assessments
* Body Mass Index (BMI) of ≥18 to ≤30 kg/m2 and weight of ≥50 to ≤100 kg.
* Non-fertile females

Exclusion Criteria:

* History of hypersensitivity, allergy or atopic/skin disease as judged by Investigator.
* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study as judged by the Investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
VAS, HPT | Visit 2-4

SECONDARY OUTCOMES:
eVAS, HPT, Laser Doppler imaging,WDT, Somedic allodynia | Visit 2-4
Vital signs, laboratory variables and adverse event each day throughout the study. paper printout ECG and/or digital ECG throughout the study. Pain evoked assessments visit 1-3 | Visit 1-5
Pharmacokinetics/Pharmacodynamics | Visit 2-4

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Berg, Study Chair — AstraZeneca R&D Södertälje; Ingemar Bylesjö, Principal Investigator — AstraZeneca R&D CPU Karolinska University Hospital, Stockholm